CLINICAL TRIAL: NCT05293574
Title: Randomized Control Trial Between Norethisterone Acetate and Expectant Management in Treatment of Simple Ovarian Cysts
Brief Title: A Trial of Norethisterone Acetate and Expectant Management in Treatment of Simple Ovarian Cysts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Mostafa Mohamed Swafi, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: simple ovarian cyst
Record Dates: First submitted 2022-03-01; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cyst Simple
MeSH Terms: interventions — Norethindrone Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norethisterone acetate group (Experimental): . In the norethisterone acetate group, the women will receive of norethisterone acetate 5 mg twice daily and are counseled about how to take norethisterone acetate and informed of possible side effects. They also receive a diary card for recording norethisterone acetate intake to be returned to the physician on the day of the next visit. An appointment for the women in both groups was scheduled at one month of treatment for the second ultrasonography.
  If there is no remission occurred another month of Norethisterone acetate will be given .
  Interventions: Drug: norethisterone acetate
- expectant managment group (No Intervention)

INTERVENTIONS:
Drug: norethisterone acetate — Norethindrone, a progesterone agonist
  Arms: norethisterone acetate group

SUMMARY:
To compare the effectiveness of (norethisterone acetate) in the treatment of spontaneously occurring simple ovarian cyst detected by ultrasonography compared with expectant management.

DETAILED DESCRIPTION:
An ovarian cyst is a sac filled with liquid or semiliquid material that arises in an ovary. The number of diagnoses of ovarian cysts has increased with the widespread implementation of regular physical examinations and ultrasonographic technology.

The discovery of an ovarian cyst causes considerable anxiety in women who fears of malignancy, but the majority of ovarian cysts are benign.

These cysts can develop in females at any stage of life, from the neonatal period to postmenopause. Most ovarian cysts, occur during adolescence, which are hormonally active periods of development.

Most are functional in nature and some times resolve without treatment. However, ovarian cysts can herald an underlying malignant process or, possibly, distract the clinician from a more dangerous condition, such as ectopic pregnancy, ovarian torsion, or appendicitis.

When ovarian cysts are large, persistent, painful, or have concerning radiographic or exam findings, surgery may be required, sometimes resulting in removal of the ovary. If a cyst does not resolve after several menstrual cycles, it is unlikely to be a functional cyst, and further workup is indicated.

Early epidemiological studies reported an inverse relationship between use of oral contraceptives (OCs) and surgically confirmed functional cysts . Many previous studies have indicated that the use of Oral Contraceptive pills (OC) is associated with a lower risk of occurrence of functional ovarian cysts. few studies have considered the treatment effect of OC on functional ovarian cysts. In current clinical practice, gynecologists treat functional ovarian cysts with either OC or expectant management alone. Several randomized controlled trials have shown no significant difference in the resolution of functional ovarian cysts treated with OC over expectant management alone Functional ovarian cyst can occur due to estrogen hyperstimulaton and some theories conceoted that progesterone treatment can suppress this cyst .

ELIGIBILITY:
Inclusion Criteria:

1. women at age 24-49 years old
2. women with simple cyst.( with none of the following: solid parts, papillary formations, peritoneal masses, intraabdominal lymph node enlargement or ascites ) .(13)
3. from 5 to10cm in diameter.
4. functioning cyst.( defined as largest dimension between 2-8 cm in diameter, unilateral, uniloculated, thin-walled, anechogenic and has distal acoustic enhancement )

Exclusion Criteria:

1. premenarche
2. postmenopause
3. current user of Norethisterone acetate.
4. those having contraindication from Norethisterone use.
5. gynecologic malignancy

Ages: 24 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
randomized control trial between (norethisterone acetate)and expectant management in Treatment of simple Ovarian Cysts | baseline
  Women who had a functional ovarian cyst will be informed about the study.They are then allocated to one or other of the treatment groups (norethisterone acetate or expectant management). the women will be returned to the physician on the day of the next visit. An appointment for the women in both groups was scheduled at one month of treatment for the second ultrasonography. cysts are measured on the day that the participants visited gynecologic clinic by transvaginal or transabdominal US who serviced gynecological patients on a regular basis The following definitions of outcomes were used: Remission, the was defined as ultrasonographic examination being unable to detect the ovarian cyst; Persistence as ultrasonographic examination being able to detect the same ovarian cyst with the same size If there is no remission occurred another month of Norethisterone acetate will be given .

CONTACTS AND LOCATIONS:
Overall Officials: abobakr alsokary abbas, prof.dr, Principal Investigator — assiut

IPD SHARING:
Plan to Share IPD: Undecided